CLINICAL TRIAL: NCT03013101
Title: A Phase II, Open, Multi-center and Single Arm Study Investigating Safety and Efficacy of Recombinant Humanized Anti-PD-1 mAb for Injection in Patients With Locally Advanced or Metastatic Melanoma and Standard Treatment Failure
Brief Title: Safety and Efficacy of Recombinant Humanized Anti-PD-1 mAb for Patients With Locally Advanced or Metastatic Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Junshi-JS001-BJZL-II
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Advanced Melanoma; Metastatic Melanoma
Keywords: anti-PD-1 monoclonal antibody; advanced; metastatic; melanoma
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- humanized anti-PD-1monoclonal antibody (Experimental): humanized anti-PD-1 monoclonal antibody is to be injected intravenously 3mg/kg Q2w until disease progresses or unacceptable tolerability occurs
  Interventions: Biological: humanized anti-PD-1 monoclonal antibody toripalimab

INTERVENTIONS:
Biological: humanized anti-PD-1 monoclonal antibody toripalimab — humanized anti-PD-1 monoclonal antibody (JS001) is a programmed death-1 (PD-1) immune checkpoint inhibitor antibody, which selectively interferes with the combination of PD-1 with its ligands, PD-L1 and PD-L2, resulting in the activation of lymphocytes and elimination of malignancy theoretically.
  Other Names: JS001, TAB001

SUMMARY:
This is a multi-center, open-label, phase 2 study evaluating the humanized anti-PD-1 antibody JS001, as a monotherapy in patients with locally advanced or metastatic melanoma who have failed in routine systemic treatment.

DETAILED DESCRIPTION:
This is a multiple-center, open-label, phase 2 study evaluating the humanized anti-PD-1 antibody JS001, as a monotherapy in patients with locally advanced or metastatic melanoma who have failed in previous routine systemic treatment. Patients are injected with JS001 with 3mg/kg every 2 weeks until disease progresses or unacceptable toxicity occurs. Response assessment is conducted by every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female aged 18 and older are eligible;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
* Histologic diagnosis of locally advanced or metastatic melanoma, while ocular melanoma is excluded, and the overall rate of mucousal melanoma is no more than 25%.
* Have failed at least 1 prior routine regimen for advanced disease.
* Providing with tumor specimen (for testing the expression of PD -L1 and the infiltrating lymphocytes);
* documentary evidence of BRAF mutation status;
* At least 1 measurable lesion (only 1 measurable lymph node lesion is excluded) (routine CT scan >=20mm, spiral CT scan >=10mm, no prior radiation to measurable lesions) Predicted survival >=3 months;
* Brain or meningeal metastases must be disposed with surgery or radiation, and be stable clinically for at least 3 months (prior systemic steroids was allowed, but concurrent administration of systemic steroids with the study drug is excluded).
* Screening laboratory values must meet the following criteria（within past 14 days）:

hemoglobin ≥ 9.0 g/dL; neutrophils ≥ 1500 cells/ µL; platelets ≥ 100 x 10^3/ µL; total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; serum creatinine ≤1╳ULN，creatinine clearance >50ml/min (Cockcroft-Gault equation) PT/INR, aPTT≤1.5 x ULN;

* Without systemic steroids within past 4 weeks
* Males or female of childbearing potential must: agree to use using a reliable form of contraception (eg, oral contraceptives, intrauterine device, control sex desire, double barrier method of condom and spermicidal) during the treatment period and for at least 12 months after the last dose of study drug.
* Must have read, understood, and provided written informed consent voluntarily. Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Prior treatment with anti-PD-1/PD-L1/PD-L2 antibody;
* Hypersensitivity to recombinant humanized anti-PD-1 monoclonal Ab or its components.
* Prior treatment with mAb within past 4 weeks.
* Prior antitumor therapy (including corticosteroids and immunotherapy) or participation in other clinical trials within past 4 weeks, or have not recovered from toxicities since the last treatment;
* Pregnant or nursing;
* Positive tests for HIV, HCV, HBsAg or HBcAb with positive test for HBV DNA (>500IU/ml)
* History with tuberculosis;
* Patients with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism or hypothyroidism.
* Severe, uncontrolled medical condition that would affect patients' compliance or obscure the interpretation of toxicity determination or adverse events, including active severe infection, uncontrolled diabetes, angiocardiopathy (heart failure > class II NYHA, heart block >II grade, myocardial infarction, unstable arrhythmia or unstable angina within past 6 months, cerebral infarction within past 3 months) or pulmonary disease ( interstitial pneumonia, obstructive pulmonary disease or symptomatic bronchospasm).
* Evidence with active CNS disease.
* meningeal carcinomatosis;
* Prior treatment with bone marrow stimulating factors，such as CSF (colony stimulating factor), EPO (erythropoietin), within past 2 weeks
* Prior live vaccine therapy within past 4 weeks.
* Prior major surgery within past 4 weeks (diagnostic surgery excluded).
* Psychiatric medicines abuse without withdrawal, or history of psychiatric illness.
* Prior malignancy active within the previous 5 years except for locally curable cancers that have been apparently cured, such as basal cell skin cancer or carcinoma in situ of the cervix.
* Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2018-09-16 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 and irRECIST Objective response rate (ORR) by RECIST 1.1 and irRECIST | 3 years

SECONDARY OUTCOMES:
Duration of response (DOR) by RECIST1.1 and irRECIST | 3 years
Progression free survival (PFS) by RECIST1.1 and irRECIST | 3 years
Overall survival (OS) | 3 years
Immunogenicity of anti-PD-1 monoclonal antibody | 1.5 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1.5 years

OTHER OUTCOMES:
Correlation analysis of PD-L1 expression of tumor by Immunohistochemistry and ORR | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, PhD, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (6):
- China (6):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer center, Guangzhou, Guangdong
  - Wuhan Union Hospital, Wuhan, Hubei
  - The 81st Hospital of Chinese People's Liberation Army, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Yunnan Cancer Hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Topalian SL, Sznol M, McDermott DF, Kluger HM, Carvajal RD, Sharfman WH, Brahmer JR, Lawrence DP, Atkins MB, Powderly JD, Leming PD, Lipson EJ, Puzanov I, Smith DC, Taube JM, Wigginton JM, Kollia GD, Gupta A, Pardoll DM, Sosman JA, Hodi FS. Survival, durable tumor remission, and long-term safety in patients with advanced melanoma receiving nivolumab. J Clin Oncol. 2014 Apr 1;32(10):1020-30. doi: 10.1200/JCO.2013.53.0105. Epub 2014 Mar 3. PMID 24590637